CLINICAL TRIAL: NCT05143255
Title: Developing a Communication Intervention to Help People With Memory Challenges and Their Care Partners Engage in Advance Care Planning
Brief Title: Developing a Communication Intervention for People With Memory Challenges and Their Care Partners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-04023598; R21AG070501 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2021-12-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Dementia
Keywords: caregiving; advance care planning; communication
MeSH Terms: conditions — Alzheimer Disease; Dementia; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KNOW Intervention (Experimental)
  Interventions: Behavioral: KNOW

INTERVENTIONS:
Behavioral: KNOW — KNow the Optimal Way (KNOW) is a manualized ADRD patient-care partner intervention designed to increase engagement in advance care planning (ACP) and completion of advance directives among early stage ADRD patients and their care partners using theoretically grounded distress tolerance techniques (inhibitory learning theory) and communication skills (cognitive-social processing theory) consistent with recommended guidelines for discussions about ACP in ADRD care.

SUMMARY:
The proposed research is consistent with broader public health goals focused on improving communication regarding end-of-life care and the Centers for Medicare and Medicaid Services' (CMS) call for increased patient engagement in advance care planning (ACP) as part of standard care. The proposed study will address this public health issue by developing a communication-based intervention designed to improve Alzheimer's Disease and Related Dementias (ADRD) patients' and care partners' engagement in ACP, distress and care partner burden, and completion of advance directives and receipt of goal-concordant care at the end-of-life. Therefore, this study is aligned with the National Institute on Aging's long-term goal to improve the quality of care for ADRD patients and CMS's goal to increase engagement in ACP.

DETAILED DESCRIPTION:
The goals of this study are to: (1) develop a communication-based intervention, called KNow the Optimal Way (KNOW) for Alzheimer's Disease and Related Dementias (ADRD) patients and care partners that includes theoretically grounded communication strategies (e.g., acknowledgment, validation of fears) and distress management techniques (e.g., deep breathing, muscle relaxation); (2) evaluate the feasibility and acceptability of the intervention; and (3) test the preliminary efficacy of the intervention on ADRD patients' and care partners' preparedness for and engagement in advance care planning (ACP), and completion of advance directives (primary outcomes) as well as patient-care partner concordance on the person with dementia (PWD)'s healthcare values, perceived need for ACP, psychological distress, communication quality, and care partner burden (secondary outcomes).

ELIGIBILITY:
Patient/care recipient (CR) eligibility criteria:

1. Montreal Cognitive Assessment-Blind (MoCA-B) score of 9-18;
2. decision-making capacity to consent to a low risk study as indicated by a score of ≥9 on the University of California-San Diego Brief Assessment of Capacity to Consent, a 10-item measure validated in patients with challenges in memory;
3. capacity to execute a Health Care Proxy, as indicated by a score of ≥ 11 on the validated and reliable HCP Guidelines for ability to execute a HCP among nursing home residents;
4. age ≥ 65;
5. reports receiving care and/or support from an unpaid care partner; and
6. reports that at least one of their ADs has not been completed (for CR's enrolled without a CP only).

Care partner (CP) eligibility criteria:

1. provides informal (unpaid) care for a person with memory challenges, per self-report;
2. MoCA-B score of ≥19; and reports that at least one of the CR's ADs has not been completed (for CPs enrolled without a patient only). While care partners must report caring for a person with memory challenges, the care partner can be enrolled in the study even if the patient is not enrolled.

Eligibility criteria for CRs and CPs enrolled as a dyad: In addition to the criteria above for CR and CP: (1) the CR and/or CP report that at least one of the CR's ADs has not been completed.

Patient and care partner exclusion criteria:

1. not fluent in English;
2. ≤17 years of age;
3. too ill or weak to complete the interviews (per the interviewer);
4. presence of significant sensory, language, or motor deficit (e.g., visual or hearing loss, paralysis, aphasia) (per self report, the interviewer or medical record); or
5. patient is in the late stage of dementia (i.e., severe cognitive impairment), is bed-bound, or has a nursing home admission planned within 12 months per CP report or the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in advance care planning preparedness, as measured by the Advance Care Planning Engagement Survey: Process Measures | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Change in advance care planning preparedness will be assessed in patients and care partners using the reliable and valid Advance Care Planning Engagement Survey: Process Measures (31-items). Response options range from 1=never to 5=a lot. Questions include those asking about knowledge of advance care planning, degree of contemplation about advance care planning, and self-efficacy and readiness to engage in advance care planning. Overall scores can range from 31 to 155, with higher scores indicating more engagement in advance care planning.
Change in patients' engagement in advance care planning, as measured by the Decision Maker subscale of the Advance Care Planning Engagement Survey: Action Measures | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Change in patient engagement in advance care planning will be assessed in patients using the reliable and valid Decision Maker (four items) subscale of the Advance Care Planning Engagement Survey: Action Measures. Response options range from 1=never to 5= a lot. Questions include those asking about whether patients have engaged in a decision around advance care planning (e.g., "Have you already decided who you want your medical decision maker to be?" Scores can range from 4 to 20, with higher scores indicating that more decisions have been made around advance care planning.
Change in care partners' engagement in advance care planning, as measured by the Van Scoy and Sudore measure which adapts the Decision Maker subscale of the Advance Care Planning Engagement Survey | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Change in care partner engagement in advance care planning will be assessed with a companion measure in the final phases of validation by Van Scoy and Sudore. This measure adapts the Advance Care Planning Engagement Survey to apply to care partners. Response options range from 1=never to 5=a lot. Scores can range from 4 to 20, with higher scores indicating more decisions have been made.
Change in discussion of advance directives | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Discussion of advance directives will be assessed with an 8-item measure that asks persons with ADRD and care partner whether the patient has discussed end-of-life care, living will, health care proxy, and DNR orders with family/patient and doctor/patient's doctor. Response options are yes or no. A total score is created by adding up the number of discussions, which can range from 0 to 8, with 0 meaning no discussions have occurred (low score) to 8, meaning all discussions have occurred (high score).
Change in the number of patients who have completed advance directives | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Completion of advance directives will be assessed by asking patients whether they have completed a do-not-resuscitate order, a living will, and/or or identified a health care proxy; data will be verified through the patient's electronic health record. Completion will be scored a 0 if the patient has completed none and 1 if they have completed one or more of the advance directives. Additional analyses will be done on each individual advance directive (e.g., 0 if no DNR order, 1 if yes to completing DNR order).

SECONDARY OUTCOMES:
Change in concordance on healthcare values, as measured by the Health Care Values Rating Scale | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Change in concordance on healthcare values will be assessed by ADRD patients' and care partners' ratings of the ADRD patient's values on the Health Care Values Rating Scale, a 13-item measure of the degree to which various values influence medical treatment decisions developed in ADRD patients. Each item is rated on a three-point Likert scale (1=influence not at all to 3=influence a lot). Concordance will be defined as a difference of one or less per item between responses of ADRD patients and their care partners (rating the ADRD patient's values).
Change in perceived need for advanced care planning (ACP), as measured by the Decisional Balance scale | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Change in perceived need for advance care planning will be assessed with the reliable and validated Decisional Balance scale, a 12-item scale that assesses perceived pros and cons of engaging in ACP. Each item is rated on a five-point Likert scale (1=not important to 5=extremely important) indicating how important a certain feature of advance care planning is. Overall scores can range from 12 (low importance) to 60 (high importance).
Change in psychological distress/depression, as measured by the Center for Epidemiological Studies Depression Scale | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Change in psychological distress will be assessed with the 20-item Center for Epidemiological Studies Depression Scale which has demonstrated validity in ADRD patients and their care partners and the seven-item anxiety subscale of the Hospital Anxiety and Depression Scale. Each item rates the degree of occurrence of certain depressive features from rarely or none of the time (less than 1 day) to most or all of the time (5-7 days). Total scores can range from 20 to 80, with higher scores indicating higher frequency.
Change in psychological distress, as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Psychological distress will be measured using the Hospital Anxiety and Depression Scale (HADS), a valid and reliable 14-item, Likert-type self-report measure of mood disturbance commonly used with cancer patients. The HADS contains two seven-item subscales: 1) anxiety and 2) depressive symptoms. Each item on this scale is rated on a 4-point scale (0 to 3), and all items are summed to create a HADS total score. Total scores can range from 0 to 42, with higher numbers indicating higher levels of distress.
Change in communication quality, as measured by the Family Communication Subscale of the Cancer Communication Assessment Tool for Patients and Families (CCAT-PF) | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Communication quality will be assessed with the 5-item Family Communication subscale of the Cancer Communication Assessment Tool for Patients and Families, a valid measure in cancer patients and care partners. Response options are on a 5-point Likert-type scale (1 = strongly disagree to 5= strongly agree). Scores can range from 5 to 25, with higher scores indicating worse communication quality.
Change in care partner burden (care partner only), as measured by the Zarit Burden Interview | Baseline, Post-Intervention (within 2 weeks), 3-month follow up
  Care partner burden will be assessed with the Zarit Burden Interview (ZBI), a reliable and valid 22-item measure of caregiver (care partner) burden used in intervention studies of cancer caregivers (care partners). Response options are on a 5-point Likert-type scale (0 = never to 4=nearly always). Scores can range from 0 to 88, with higher scores indicating higher levels of burden.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Czaja, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No